CLINICAL TRIAL: NCT01576276
Title: A Brain Imaging Study of Opioid (Morphine) and Non-opioid (Ketorolac) Conditioning Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2011P000358
Record Dates: First submitted 2012-02-24; First posted 2012-04-12 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Healthy Controls
MeSH Terms: interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine condition (Experimental)
  Interventions: Radiation: Integrated MR-PET scan
- Ketorolac condition (Experimental)
  Interventions: Radiation: Integrated MR-PET scan; Drug: Ketorolac

INTERVENTIONS:
Radiation: Integrated MR-PET scan — Integrated MR-PET scan using [11C]diprenorphine
Drug: Ketorolac — 3 administrations of ketorolac over course of study
  Arms: Ketorolac condition

SUMMARY:
Healthy right-handed volunteers aged 21 to 50 needed for a research study of the effects of morphine and ketorolac on brain activity in response to pain stimuli as measured by functional Magnetic Resonance Imaging (fMRI) and Positron Emission Tomography (PET). Study will be conducted on six separate days not requiring an overnight stay in the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female adults, aged 21-50
2. No contraindications to fMRI scanning
3. Within 15% of normal BMI
4. Right handed (dominant hand is right hand)
5. Have taken an opioid drug at least once in the past (for example, after a surgery)

Exclusion Criteria:

1. Current or past history of major medical, neurological, or psychiatric illness
2. Women who are pregnant or breast feeding, have gone through menopause, or have irregular menstrual cycles (length of cycle must be within 26 to 32 days)
3. Contraindications to morphine administration:

   * i) Hypersensitivity to morphine or other phenanthrene-derivative opioid agonists (codeine, oxycodone, etc.), morphine salts, or any component of the product
   * ii) Concomitant use of other CNS depressants including antihistamines or alcohol
   * iii) History of drug or alcohol abuse
   * iv) History of head trauma
   * v) History of liver problems
   * vi) Pre-existing respiratory conditions (ex. COPD, asthma)
   * vii) Current use of any drugs that interact with morphine
4. Contraindications to ketorolac administration

   * i) Allergic-type reaction, or urticaria in response to exposure to aspirin or other NSAIDS
   * ii) Concomitant aspirin or NSAID use
   * iii) Hypersensitivity previously demonstrated to ketorolac tromethamine or to any product component
   * iv) Peptic ulcer disease (active or history), or other gastrointestinal problems
   * vi) Current use of any drugs that interact with ketorolac (ex. heparin/warfarin)
   * vii) History of bleeding disorder
   * viii) Low body weight, under 50 kg
5. Contraindications to fMRI scanning (including cardiac pacemaker, metal implants, claustrophobia, pregnancy)
6. Contraindications to either of the emergency medications (Ondansetron or Narcan)
7. History of head trauma
8. High blood pressure (>140 systolic, >90 diastolic)
9. History of impaired urinary elimination
10. Major kidney problems, bleeding problems, severe dehydration, or recovering from a recent surgery (within past year).
11. Instability of responses to experimental pain (see Study Procedures Section)
12. History of asthma
13. History of diabetes
14. Liver Function Test results greater than 2.5 times the upper limit of normal (ULN) at Screening
15. History of smoking (past or current)
16. Use of psychotropic drugs, hormone treatments (including hormonal birth control) within 1 year
17. Non-fluent speaker of English
18. Positive urine drug screen (i.e. positive on any of the 10 measures tested, including cocaine, marijuana, opiates, amphetamines, methamphetamines, phencyclidine, barbiturates, benzodiazepines, methadone, and tricyclic antidepressants)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Morphine Condition: Integrated MR-PET scan: Integrated MR-PET scan using [11C]diprenorphine
  Morphine: 3 administrations of morphine over course of study
Period: Overall Study
Arm/Group | Morphine Condition | Ketorolac Condition
Started | 22 | 29
Completed | 14 | 18
Not Completed | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine Condition | Ketorolac Condition | Total
Number analyzed (Participants) | 22 | 29 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (3.3) | 26.0 (4.9) | 25.5 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 17 | 22 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 19 | 26 | 45
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 23 | 41
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 1 | 1
Pain Ratings [Mean (Standard Deviation); unit: scores on a scale] — Population: Some subjects were dropped before or during the MRI scan in which baseline pain ratings were collected. We used the Gracely Sensory Pain Scale (0-20; 0: no pain, 20: intolerable pain) to rate the pain subject's experienced.
  scores on a scale
    number analyzed (Participants) | 14 | 18 | 32
    (all) | 10.9 (2.6) | 11.6 (2.2) | 11.3 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: fMRI Signal Changes
Description: Obtain information about brain activity, including BOLD (Blood-oxygen-level dependent) signal, using an fMRI system. Data analysis was applied using SPM 12 with a standard pipeline.
Time Frame: one day
Population: Here we present the average fMRI (functional MRI) signal changes of clusters that survived a threshold of 0.005 with10 continuous voxels. We only reported beta values in pain related areas.
Measure: Mean (Standard Deviation); unit: Beta value
Groups:
- fMRI Signal Change: We used SPM 12 to analyze the data, and compared the fMRI signal change during pressure pain between 1. morphine injection cue vs. control cue, 2. ketorolac injection cue vs. control cue. A threshold of p < 0.005 with 10 continuous voxels was applied.
Arm/Group | fMRI Signal Change
Number analyzed (Participants) | 33
Beta value
  morphine injection cue at operculum | 0.82 (0.79)
  morphine control cue at operculum | 0.43 (0.65)
  ketorolac injection cue at operculum | -0.02 (0.46)
  ketorolac control cue at operculum | 0.55 (0.53)
  ketorolac injection cue at insula | 0.09 (0.42)
  ketorolac control cue at insula | 0.85 (0.92)

2. Primary Outcome: Pain Ratings
Description: The primary endpoint was the morphine and ketorolac conditioning effects as indicated by subjective pain rating changes between pain only (a control condition with no injection of glucose, but subject's did see an image of an hour glass displaying how much time they had before receiving a painful stimulus) and pain+glucose (subjects received a glucose injection accompanied by an injection schematic followed by a painful stimulus) within the morphine and ketorolac groups. We used the Gracely pain rating scale (ranging from 0, no sensation to 20, extremely painful).
Time Frame: One day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Morphine Condition | Ketorolac Condition
Number analyzed (Participants) | 14 | 18
units on a scale | -0.22 (1.45) | -0.97 (2.81)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant over a 3 hours period (from time of drug administration until they left 3 hours later). We collected this for every participant throughout our study.
Description: Our definitions are consistent. After every drug administration we asked a standard questionnaire, which we also asked again a couple of hours following the initial drug administration. Specifically, we asked subjects if they felt nauseous, indigestion, itching, spacey/drugged, lightheadedness/faint, sense of difficulty concentrating, or sleepy.
Arm/Group | Morphine Condition | Ketorolac Condition
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/29
Other Adverse Events (participants affected / at risk) | 5/22 | 1/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine Condition (N=22) | Ketorolac Condition (N=29)
Drug related reactions (Surgical and medical procedures) | 5 (5) | 1 (1) — Drug related reactions to morphine and ketorolac, including feeling nauseous, spacey, and drugged.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT01576276/Prot_SAP_000.pdf